CLINICAL TRIAL: NCT02607397
Title: In Silico Clinical Trial on Irradiation Low Grade Glioma, Comparing Photon and Proton Therapy: A Multicentric Planning Study Based on a Reference Dataset of Patients
Brief Title: ROCOCO - Low Grade Glioma - Planning Study
Acronym: ROCOCO LGG
Status: Completed | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Collaborators: University Medical Center Nijmegen (Other); Radiotherapy Group Deventer (Other); Heidelberg University (Other); University of Giessen (Other)
Responsible Party: Sponsor
Other Study IDs: ROCOCO LGG
Record Dates: First submitted 2015-11-12; First posted 2015-11-18 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Low Grade Glioma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The cost of particle therapy (PT) are considerably higher than conventional radiotherapy (RT) with photons. Considering potential dosimetric advantages of PT, it is necessary to determine if PT are more cost-effective than photons per indication regarding quality of life, survival, and progression free survival. Given the lack of evidence for the benefit of particle therapy in relevant cases, investigators proposed an in silico trial to investigate to what extend proton therapy decrease the amount of irradiated normal tissue and, consequently, the risk of side effects in the surrounding normal tissue as well as the risk of secondary tumors. Given validated dose-response curves and/or NTCP models, a 10% lower mean dose of proton therapy on normal tissue compared to photon therapy should result in at least a 20% lower risk of side effects.

DETAILED DESCRIPTION:
Patients with low grade glioma have a far better prognosis than patients with high grade glioma. Despite their low incidence and initial favorable biological behavior, low-grade gliomas are behaving as malignant brain tumours leading to considerable morbidity and mortality especially in young patients. Low-grade infiltrating gliomas in adults include diffuse astrocytoma, oligoastrocytoma and oligodendroglioma. With the WHO 2007 classification the variety within the low grade glioma patient group was large. With the introduction of molecular marker like IDH, MGMT, 1p/19q the classification of glioma's in general is a matter of debate, because shifts in treatments and prognosis. In this context, the importance of molecular markers is recognized and used for designing new trials.

Because of this improved determining of long term survivors like low grade glioma patients, reducing the long term side effect becomes even more relevant. One of the prominent side effect of radiotherapy in low grade glioma patients is the decline in neurocognitive function and loss of memory. This enables patients in their daily activities and causes loss of quality of life. The hippocampus and associated limbic system have long been known to be important in memory formation and pre-clinical models show loss of hippocampal stem cells with radiation as well as changes in architecture and function of mature neurons. Cognitive outcomes in clinical studies are beginning to provide evidence of cognitive effects associated with hippocampal dose and the cognitive benefits of hippocampal sparing. With currently developing IMRT techniques attempts are made to lower the dose to the hippocampus. Besides the hippocampus the dose to the posterior part of the cerebellum seems to influence cognition. Koziol wrote recently the current consensus paper which gathers diverse views on a variety of important roles played by the cerebellum across a range of cognitive and emotional functions. This paper considers the cerebellum in relation to neurocognitive development, language function, working memory, executive function, and the development of cerebellar internal control models and reflects upon some of the ways in which better understanding the cerebellum's status as a "supervised learning machine" can enrich our ability to understand human function and adaptation.

This in silico planning study compares different treatments (photon, proton and C-ion) focusing on normal tissue radiation exposure for a fixed tumor dose, using the same delineation of gross target volume (GTV), clinical target volume (CTV) and planning target volume (PTV). The comparison will be based on dosimetric parameters on normal tissues such as mean hippocampus dose, etc. In addition, the NTCP for a fixed tumor dose or the same expected TCP will be determined. Cobalt Gy equivalent doses will be used when reporting the proton and C-ion dose. In the case of protons, a constant RBE value of 1.1 will be used for both the tumor and the normal tissues. The RBE of C-ions will be calculated based on the models used by the participating centers. The GSI in-house treatment planning system uses RBE values calculated on the basis of the local effect model (LEM). The LEM I (alpha/beta=2) is based on the radial dose distribution of each charged particle crossing into a cell nucleus, as well as on the radiosensitivity and repair capacity of the tissue. The TPSs used by UHM is also based on the LEM model. The model used at NIRS utilizes fixed RBE values that are dependent on the depth in the body, but independent of dose level or tumor type.

ELIGIBILITY:
Inclusion Criteria:

* Low Grade Glioma patients
* Treated with radical intent

Exclusion Criteria:

* No Low Grade Glioma

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 25 patients. Each patient will function as his or her own control.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2015-05; Primary Completion 2017-03 (Actual); Study Completion 2017-03 (Actual)

PRIMARY OUTCOMES:
Dmean | 1 month
  The normal tissue dose volume parameters per tumor type are defined as Hippocampus: Dmean
Dmax | 1 month
  The normal tissue dose volume parameters per tumor type are defined as Hippocampus: Dmax

SECONDARY OUTCOMES:
Normal Tissue Complication Probability | 1 month
  Based on the OAR's radiation exposure, normal tissue complication probability (NTCP) will be calculated using existing models or existing dose response curves.

CONTACTS AND LOCATIONS:
Overall Officials: Philippe Lambin, MD, PhD, Principal Investigator — Maastro Clinic, The Netherlands
Locations (4):
- Germany (2):
  - University of Heidelberg, Heidelberg
  - University Hospital Giessen and Marburg, Marburg
- Netherlands (2):
  - Radiotherapy Group, Deventer
  - University Medical Center Nijmegen, Nijmegen